CLINICAL TRIAL: NCT02846818
Title: Continuous Monitoring of Cerebral Energy State During Cardiac Surgery - A Novel Approach Utilizing Intravenous Microdialysis
Brief Title: Cerebral Energy State in Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Simon Mölström, MD, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: S-20130166
Record Dates: First submitted 2016-07-19; First posted 2016-07-27 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Postoperative; Dysfunction Following Cardiac Surgery
Keywords: Microdialysis; Cardiac surgery; Lactate to pyruvate ratio; Cardiopulmonary bypass; Neurological complications
MeSH Terms: interventions — Microdialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low mean arterial perfusion pressure (Experimental): 5 patients undergoing primary, elective coronary artery bypass grafting were randomized to usual range MAP (40 to 60 mmHg) during CPB. Microdialysis catheters were positioned in a retrograde direction in the internal jugular vein.
  Interventions: Procedure: Microdialysis
- High mean arterial perfusion pressure (Experimental): 5 patients undergoing primary, elective coronary artery bypass grafting were blindly randomized to intervention group MAP (60 to 80 mmHg) during CPB. Microdialysis catheters were positioned in a retrograde direction in the internal jugular vein.
  Interventions: Procedure: Microdialysis

INTERVENTIONS:
Procedure: Microdialysis — Extracerebral MD catheters were positioned in a retrograde direction in the internal jugular vein.
  Other Names: MMSE; NIRS

SUMMARY:
Impaired cerebral function remains an important complication of cardiopulmonary bypass (CPB) during cardiac surgery. The aim of the present study is to investigate whether the lactate to pyruvate (LP) ratio obtained by microdialysis (MD) of the cerebral venous outflow reflects a derangement of global cerebral energy state during cardiopulmonary bypass.

DETAILED DESCRIPTION:
Patients undergoing primary, elective coronary artery bypass grafting were blindly randomized to usual range MAP (40 to 60 mmHg; n = 5) or intervention group MAP (60 to 80 mmHg; n = 5) during CPB. MD catheters were positioned in a retrograde direction in the internal jugular vein and a reference catheter was inserted into the brachial artery. The relations between LP ratio, MAP, data obtained from bi-frontal NIRS and neurological outcome measures were assessed.

ELIGIBILITY:
Inclusion criteria:

* Elective CABG on CPB

Exclusion criteria:

* Acute patients or reoperations
* Patients with epidural catheter
* Previous stroke
* Stenotic carotids
* Ejection fraction (EF) < 50 %
* Estimated per operative risk > 5%

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-02; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Extracerebral microdialysis parameters | MD parameters were measured intraoperatively and for two hours postoperatively
  Does the LP ratio of cerebral venous blood increase significantly during CPB indicating compromised cerebral oxidative metabolism.The analyses included the variables routinely monitored during intracerebral microdialysis: glucose, pyruvate, lactate, glutamate, glycerol and lactate to pyruvate ratio.

SECONDARY OUTCOMES:
Mini mental state examination (MMSE) | Neurological complications with in 2 days after surgery
  Patients were assessed preoperatively and postoperatively day two after surgery
Near-infrared spectroscopy (NIRS) | one day
  Right and left frontal rSO2 values were recorded simultaneously pre- and intraoperatively and for two hours postoperatively. Cerebral desaturation was defined as a decrease in the relative rSO2 value of 20 % compared with the individual pre-induction baseline value

CONTACTS AND LOCATIONS:
Overall Officials: Palle Toft, Professor, Study Director — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Fyn, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Background] Ahonen J, Salmenpera M. Brain injury after adult cardiac surgery. Acta Anaesthesiol Scand. 2004 Jan;48(1):4-19. doi: 10.1111/j.1399-6576.2004.00275.x. PMID 14674968
- [Background] McDonagh DL, Berger M, Mathew JP, Graffagnino C, Milano CA, Newman MF. Neurological complications of cardiac surgery. Lancet Neurol. 2014 May;13(5):490-502. doi: 10.1016/S1474-4422(14)70004-3. Epub 2014 Apr 2. PMID 24703207